CLINICAL TRIAL: NCT06025656
Title: Assessment of the Reliability and Validity of the Leg Lateral Reach Test to Measure Thoraco-Lumbo-Pelvic Rotation in Adolescent Tennis Players
Brief Title: Assessment of the Reliability and Validity of the Leg Lateral Reach Test in Adolescent Tennis Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Sevim Beyza Ölmez, Principal Investigator, Gazi University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-942
Record Dates: First submitted 2023-08-29; First posted 2023-09-06 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Trunk Injury; Mobility Limitation; Spine Injury; Athletic Injuries
Keywords: Spine; Leg lateral reach test; Range of motion; Tennis player; Low Back Pain; Mobility
MeSH Terms: conditions — Mobility Limitation; Spinal Injuries; Athletic Injuries; Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Other): adolescent tennis player
  Interventions: Diagnostic Test: Leg Lateral Reach Test

INTERVENTIONS:
Diagnostic Test: Leg Lateral Reach Test — To conduct the leg reach test, participants began by positioning themselves with their arms hanging at their sides. They were then guided to raise the leg under assessment and extend it across the opposite leg to make contact with a wooden bar, employing trunk rotation in the process. During each trial, participants were consistently motivated to ensure that both shoulders remained in contact with the floor and to stretch their tested leg as far as they could along the length of the wooden bar. If a participant was unable to sustain contact between their foot and the wooden bar for a duration of 5 seconds at the point of maximal reach, or if both shoulders lifted off the floor, that specific trial was considered invalid and not included in the analysis.
  Each participant completed three repetitions of this test for both the right and left sides, and the average of their reach distances was subsequently calculated for assessment.

SUMMARY:
The aim of this study is to evaluate the reliability and validity of the Leg Lateral Reach Test to measure thoraco-lumbo-pelvic segment mobility in adolescent tennis players. The fact that the test is valid and reliable for tennis players will contribute to monitoring trunk rotation flexibility in athletes, comparing them bilaterally, and revealing the exercise training necessary to improve performance.

DETAILED DESCRIPTION:
Tennis is a sport characterized by coordinated, repetitive, and rotational movements along the kinetic chain. Ineffective use of the trunk segment to generate rotational momentum is thought to increase the load on the upper extremity. Limited trunk rotation flexibility can cause abnormal trunk motion patterns, resulting in lower back injuries and pain as well as upper extremity injuries in throwing athletes. Therefore, assessment of trunk flexibility in athletes who perform repetitive trunk rotations, such as tennis players, is critical for effective rehabilitation and prevention of sports injuries.

The Leg Lateral Reach Test was developed to measure the rotation of the thoraco-lumbo-pelvic segment and was found to be valid and reliable in physically active, healthy individuals. Therefore, the aim of this study is to evaluate the reliability and validity of the Leg Lateral Reach Test to measure thoraco-lumbo-pelvic segment mobility in adolescent tennis players. The fact that the test is valid and reliable for tennis players will contribute to monitoring trunk rotation flexibility in athletes, comparing them bilaterally, and revealing the exercise training necessary to improve performance.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent tennis players

Exclusion Criteria:

* Athletes with a history of musculoskeletal injury or surgery in the last year that would prevent the tests from being performed
* Athletes who feel pain in the trunk and lower extremities during the tests

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Leg Lateral Reach Test-1 | first day
  The leg lateral reach test will be measured by the first investigator.
Leg Lateral Reach Test-2 | first day
  The leg lateral reach test will be measured by the second investigator.
Leg Lateral Reach Test-3 | 5-7 days after
  The leg lateral reach test will be measured by the first investigator.
Leg Lateral Reach Test-4 | 5-7 days after
  The leg lateral reach test will be measured by the second investigator.
Seated Rotation Test | first day
  A seated rotation test will be measured for validity analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Hazar, Study Director — Gazi University; Elif Aygün Polat, Principal Investigator — Gazi University; Sevim Beyza Ölmez, Principal Investigator — Gazi University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Result] Pontes-Silva A, Avila MA, de Araujo ADS, Penha TFC, Takahasi HY, Bassi-Dibai D, Dibai-Filho AV. Assessment of the Reliability of the Leg Lateral Reach Test to Measure Thoraco-Lumbo-Pelvic Rotation in Individuals With Chronic Low Back Pain. J Manipulative Physiol Ther. 2021 Sep;44(7):566-572. doi: 10.1016/j.jmpt.2021.12.001. PMID 35282857
- [Result] Kim SH, Kwon OY, Park KN, Hwang UJ. Leg lateral reach test: The reliability and correlation with thoraco-lumbo-pelvic rotation range. J Sci Med Sport. 2017 Jan;20(1):2-5. doi: 10.1016/j.jsams.2016.04.006. Epub 2016 May 2. PMID 27210501